CLINICAL TRIAL: NCT00035152
Title: A Multicenter, Randomized Trial for Stage IIIB or IV NSCLC Comparing Weekly Taxol(Paclitaxel) and Carboplatin(Paraplatin) Regimen Versus Standard Taxol and Carboplatin Administered Every Three Weeks, Followed by Weekly Taxol.
Brief Title: Study Comparing Weekly Taxol and Carboplatin vs Standard Taxol and Carboplatin Regimen for Stage IIIB or IV Non-Small-Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BMS TAX/MEN.12
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Carboplatin

INTERVENTIONS:
Drug: Paclitaxel and carboplatin

SUMMARY:
Taxol and carboplatin are commonly used drugs for the treatment of stage IIIB or IV non small cell lung carcinoma.

This study compares treatment with Taxol/carboplatin given every 3 weeks to a schedule where it is given weekly.

The purpose of the study is to determine the most effective and safe schedule for giving these drugs in non small cell lung carcinoma.

ELIGIBILITY:
Inclusion criteria:

* Confirmation of non-small cell bronchogenic carcinoma (epidermoid, squamous, adeno, large cell anaplastic carcinoma, but no small cell or carcinoid) must be histologically or cytologically confirmed.
* No prior antineoplastic chemotherapy, hormonal therapy or therapy with biological response modifiers
* No previous irradiation to the only area of measurable disease.

Exclusion Criteria:

* Past or current history of neoplasm other than the entry diagnosis. Exceptions are curatively treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix or other cancers treated by surgery or radiation with a disease free survival longer than 5 years.
* Patients who have undergone surgery less than 3 weeks prior to enrollment.
* History of serious cardiac disease not adequately controlled.
* Patients with serious active infections or other serious underlying medical condition.
* Uncontrolled diabetes mellitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444
Dates: Start 2000-06; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Locations (56):
- United States (56):
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Little Rock Hematology/Oncology Associates, Little Rock, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Medical Oncology Care Associates, Orange, California
  - Naval Medical Center, San Diego, California
  - Danbury Hospital/Praxair Cancer Center, Danbury, Connecticut
  - Walter Reed Army Hospital, Washington D.C., District of Columbia
  - Washington VA Medical Center, Washington D.C., District of Columbia
  - Good Samaritan Medical Center, West Palm Beach, Florida
  - Wellstar Cobb Hospital, Austell, Georgia
  - Joliet Oncology/Hematology Associates,Ltd., Joliet, Illinois
  - Mid Illinois Hematology and Oncology Associates, Ltd., Normal, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Community Cancer Care, Inc., Indianapolis, Indiana
  - Associated Physicians & Surgeons Clinic, LLC, Terre Haute, Indiana
  - Mercy Cancer Center, Mason City, Iowa
  - Siouxland Hematology/Oncology Associates, Sioux City, Iowa
  - Jewish Medical Plaza, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Louisiana Oncology Associates, Lafayette, Louisiana
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Maine General Medical Center, Waterville, Maine
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Hematology and Oncology Associates of Southern Michigan,P.C, Jackson, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Fairview-University Medical Center, University of Minnesota, Minneapolis, Minnesota
  - Metro Minnesota CCOP, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - Creighton University Cancer Center, Omaha, Nebraska
  - The Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - Hematology-Oncology of Central New Jersey, Red Bank, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Advanced Oncology Associates, Armonk, New York
  - Brooklyn VA, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Clifton Springs Hospital and Clinic, Clifton Springs, New York
  - Goshen Medical Associates, Goshen, New York
  - New York Oncology-Hematology,P.C./Capital District Hematology, Oncology Associates, Latham, New York
  - Hematology/Oncology of Rockland, New York, New York
  - Upstate New York Cancer R & E, Rochester, New York
  - Raleigh Hematology Associates, Wake Practice, Cary, North Carolina
  - Quadrangle Medical Specialists, Southern Oncology Research, Greenville, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Columbus CCOP, Columbus, Ohio
  - Central Pennsylvania Hematology & Medical Oncology Associates, P.C., Lemoyne, Pennsylvania
  - Albert Einstein Healthcare Network, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center/University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Guthrie Clinic Ltd, Sayre, Pennsylvania
  - Boston Cancer Group, PLC, Memphis, Tennessee
  - Don & Sybil Harrington Cancer Center, Amarillo, Texas
  - Brackenridge Hospital, Austin, Texas
  - Southwest Regional Cancer Center, Austin, Texas
  - Southwest Cancer Center, Lubbock, Texas
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington